CLINICAL TRIAL: NCT02225704
Title: A Phase II Study of Radium-223 in Combination With Enzalutamide in Progressive Metastatic Castrate-Resistant Prostate Cancer
Brief Title: Radium-223 in Combination With Enzalutamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL (ICORG) 13-21
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radium-223; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radium-223 and enzalutamide (Experimental): Radium-223 50kBq/kg by intravenous injection on day 1 of every 4 week cycle for maximum of 6 cycles Enzalutamide 160mg orally daily
  Interventions: Drug: Radium-223 and enzalutamide

INTERVENTIONS:
Drug: Radium-223 and enzalutamide

SUMMARY:
This study aims to determine the safety and tolerability of Radium-223 when administered in combination with enzalutamide in progressive metastatic castrate-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedures
2. Age ≥18 years and male.
3. ECOG performance status ≤ 2.
4. Histologically/cytologically confirmed adenocarcinoma of the prostate, and without neuroendocrine differentiation or small cell histology.
5. Metastatic disease as confirmed by Computed tomography (CT)/ Magnetic resonance imaging (MRI) or bone scan.
6. 6. Patients must have documented Progressive disease (PD) either by radiographic or PSA criteria as defined in a) and b) below:

   1. For the Radiographic PD assessment, 2 sets of scans using the same imaging modality (ie CT/MRI or bone scan) and taken at separate time points are required to document radiographic disease progression during or following the patient's most recent anti-neoplastic therapy, (note: the 1st bone scan can be from before most recent therapy but the 2nd scan must show disease progression during or after the most recent therapy).

      For patients with bone disease, progression will be assessed following recommendations by the Prostate Cancer Working Group (PCWG2, see Appendix FC): appearance of 2 or more new lesions on bone scan, confirmed, if necessary, by other imaging modalities (such as CT scan or MRI), if results of the bone scans are ambiguous).

      For patients with soft tissue lesions progression will be assessed using RECIST 1.1 criteria, (see Appendix GD). Patients may have measurable or non-measurable disease according to RECIST criteria version 1.1 (see Appendix GD)
   2. PSA progression is defined as an increase in PSA, as determined by 2 separate measurements taken at least 1 week apart and confirmed by a third. If the third measurement is not greater than the second measurement, then a fourth measurement must be taken and must be greater than the second measurement for the patient to be eligible for the study. Furthermore, the confirmatory PSA measurement (i.e. the third or, if applicable, fourth PSA measurement) must be defined. If a patient has received prior anti-androgen therapy (e.g. bicalutamide), PSA progression must be evident and documented after discontinuation of anti-androgen therapy, (note: The 1st PSA reading taken to document disease progression when the patient presents can be while the patient is on Casodex or other ADT).
7. Prior surgical castration or concurrent use of an agent for medical castration with testosterone at screening less than 50ng/dL.
8. Screening PSA ≥ 2 ng/mL.
9. Patients, even if surgically sterilized who (i.e. status post-vasectomy):

   * will abstain from intercourse
   * or must agree to use barrier contraception during and for 6 months after discontinuation of study treatment.
   * If the patient engages in sexual intercourse with a woman of childbearing potential, a condom and another form of birth control must be used during and for 6 months after treatment.
10. Stable medical condition
11. Life expectancy of 12 months or more based on general health and prostate cancer disease status as judged by the investigator.
12. Documented presence of osseous metastases with or without visceral involvement / lymph nodes.
13. Able to swallow study drug as whole tablet.
14. Adequate haematological, hepatic, and renal function.
15. Continuous daily use of oral prednisone, oral dexamethasone, or other systemic corticosteroids is allowed prior to study entry but must be discontinued a minimum of 2 weeks prior to start of study treatment.

Exclusion Criteria:

1. Patients should not be receiving any other investigational agents (within 30 days prior to registration)
2. Patients with Gastrointestinal (GI) tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g. Crohn's disease, ulcerative colitis).
3. Have current active hepatic or biliary disease
4. Prior therapy with orteronel, ketoconazole, aminoglutethimide, abiraterone or enzalutamide
5. All anti-androgen therapy (including bicalutamide) is excluded within 6 weeks prior to first dose of study drug. Any other therapies for prostate cancer, other than GnRH analogue therapy, such as progesterone, medroxyprogesterone, progestins (megesterol), or 5-alpha reductase inhibitors (eg, finasteride or dutasteride), must be discontinued 2 weeks before the first dose of study drug. [Bisphosphonates and Denosumab are allowed concomitant medications].
6. Prior chemotherapy for prostate cancer with the exception of:

   * neoadjuvant/ adjuvant therapy as part of initial primary treatment for local disease that was completed 2 or more years prior to screening.
   * Patients who received prior docetaxol for castrate sensitive metastatic prostate cancer commencing with 120 days of ADT initation where total dose received did not exceed 450mg/m2
7. Prior exposure to bone directed radioisotope therapy, eg samarium 153, strontium 90;
8. Exposure to external beam radiation within 4 weeks prior to receiving the first dose of study drug. In patients with untreated imminent or established spinal cord compression, treatment with standard of care, as clinically indicated, should be completed before starting treatment with Ra-223 dichloride (Xofigo®).
9. Diagnosis of or treatment for another systemic malignancy within 2 years before the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease.
10. History of myocardial infarction, unstable symptomatic ischemic heart disease/ unstable angina, uncontrolled on-going arrhythmias of Grade >2 , pulmonary embolism, or any other cardiac condition within 6 months prior to first dose of study drug.
11. New York Heart Association Class III or IV heart failure.
12. History of seizure, underlying brain injury with loss of consciousness, stroke, transient ischaemic attack (TIA), cerebral vascular accident, primary brain tumours or brain metastases, brain arteriovenous malformation, alcoholism., or the use of concomitant medications that may lower the seizure threshold.
13. Known human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C, life-threatening illness unrelated to cancer, or any ongoing serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study. Patients will be tested for hepatitis B or C or HIV infection during screening if they are considered by the investigator to be at higher risk for these infections and have not been previously tested, or if testing is required by the independent ethics committee or institutional review board.
14. Prohibited medications, including drugs that may affect exposure to enzalutamide i.e. study drugs that induce or inhibit CYP3A4, CYP2C8, and CYP2C9

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
To determine safety | approximately 6 to 9 months
  To record the incidence of grade 3 or higher adverse events during the period of combination therapy; graded according to the NCI CTCAE version 4

SECONDARY OUTCOMES:
Time to clinical and Prostate Specific Antigen (PSA) progression | Approximately 2 years
PSA response | approximately 2 years
Time to first skeletal-related event | approximately 2 years
  Time to first skeletal-related event will be analysed using the Kaplan-Meier method, presenting estimated of median PFS with 95% confidence intervals, also estimates of PFS and 95% confidence intervals at 12 months
Pain assessment | approximately 6 - 9 months
  The Brief Pain Inventory - Short Form questionnaire will be used to gather this data
Measure overall survival | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ray McDermott, Prof, Principal Investigator — St Vincent's University Hospital / AMNCH
Locations (7):
- Ireland (7):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - SLRON, St James's Hospital, Dublin
  - St Vincents University Hospital / AMNCH, Dublin
  - Tallaght Hospital, Dublin
  - Galway University Hospital, Galway